CLINICAL TRIAL: NCT06419257
Title: Investigating the Efficacy of an Augmented Virtual Reality Driving Simulator (VRDS) on Institutionalized Dementia Patients
Brief Title: Investigating the Efficacy of an Augmented Virtual Reality Driving Simulator on Institutionalized Dementia Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HS23059 (B2023:059)
Record Dates: First submitted 2023-08-01; First posted 2024-05-17 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Advance Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- VRDS users (Experimental): Individuals who would use the VRDS
  Interventions: Device: VRDS

INTERVENTIONS:
Device: VRDS — VRDS is an augmented virtual reality driving simulator.

SUMMARY:
The improvement in health and welfare in modern society has led to an increase in life expectancy. Alternatively, the longer one lives, the more likely to experience deterioration in memory, cognitive ability, and executive function skills in our brains. While some cognitive impairments can be typical results of normal aging, a decline in spatial cognition can be a sign of dementia, especially Alzheimer's disease (AD). Based on the neuroplasticity of the brain even at old ages, there are some hopes to combat dementia by repeated use of cognitive exercises in the form of a serious game designed for older adults. A popular new technology to be used to design serious games is virtual reality (VR) designs. Aside from the gaming applications, the focus of VR experiments in medicine and neuroscience is to simulate a naturalistic environment to investigate brain function and/or use it for cognitive training.

A virtual reality driving simulator (VRDS) has been developed by our team that is proposed to be installed in an existing car model at Riverview Health Center (RHC) dementia units. The VRDS has different levels of difficulty so that it can be utilized by people with different levels of cognitive impairments. However, in this study, the users will probably use only its level 1. The aim is to investigate the efficacy of the VRDS amongst institutionalized Alzheimer's/dementia patients, who are not capable of performing standard assessments. The goal is mainly to improve their mood and quality of life as many of these patients miss driving. Thus, their plausible mood change are assessed by asking the dementia unit nurses to share their observations of the patients in relation to VRDS usage; it will be a free-format anecdotal observation. In addition, while these patients are not expected to show any significant learning, playing this VRDS may improve patients' implicit memory; which can be observed by how well or poor they drive the simulated car; for example, how many times they crash to the curb or how many times they hit an animal, or how many times they ignore the red traffic light, etc.; these are reflected in the game's score.

It is anticipated that this VRDS will have an overall positive effect on users' moods, and also it may result in an implicit memory improvement.

DETAILED DESCRIPTION:
The only research instrument is the designed VRDS. Virtual Reality Driving Simulator (VRDS) Experiment The VRDS is a serious game that features three levels of difficulty and routes through a naturalistic country road. As the game progresses in each level, the route will contain various intersections. One intersection is located on the first level, while two and three intersections are located on the second and third levels. A number of traffic elements are placed along the road. Every intersection has a traffic light. There are stop signs at a few points throughout each level (one stop sign for each of the first two levels and two stop signs for the final level). In addition, an upcoming vehicle is occasionally placed in the opposite lane and during the initial stages of each level, the sudden appearance of a rural animal is simulated.

In this study, our target users are advanced stage 3 and 4 dementia (in particular Alzheimer's disease) patients who are institutionalized. Therefore, the VRDS has been designed in a way that when a participant starts using it, the game will begin from level 1. In case they successfully complete the level, then they will automatically proceed to level 2. If the game remains idle, then it will be reset to level 1. There will be no written instructions but an audio messages is played as the warning (e.g. passing a red light without stopping) and encouraging messages when they reach a target on the road.

User-specific log files are created for each training trial the user plays; they are created using an interactive input field before the training begins. Our analysis of the logged file lets us know for example whether the users have stopped at traffic signals and stop signs in a timely manner, or they have crashed to the curb, or haven't stopped when an animal jumps to the road, etc.

The VRDS will be installed in the existing car model in A-B dementia units of the RHC. The steering wheel and accelerating pedal of the car will be replaced with the steering wheel and pedals that are used as input controllers of the VRDS game. The VRDS screen on the laptop will be projected to the actual front window of the car.

In our experience, patients with advanced-stage dementia do not feel motion sickness; however, it is still possible for a participant to feel motion sickness, in that case, the research assistant next to the participant will stop the program and help the participant to get out of the car and back to their room.

ELIGIBILITY:
Inclusion Criteria:

* Living in a dementia care unit of Riverview Health Center
* Being mobile and able to see.

Exclusion Criteria:

* Residents with significant mobility issues (wheelchair users) and those with significant visual impairment will be excluded.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Nurses overall observations of the study participants on a scale of -1, 0 and 1 for worse, no change and improved, respectively. | every week for a maximum of 52 weeks
  a custom made questionnaire for interview of the nurses of the participants

SECONDARY OUTCOMES:
The Game's score through the period of the study on a value between 0 to 100 for the minimum and maximum score in the game. | every week for a maximum of 52 weeks
  The VRDS logs all the information on how the game is played. Those information is used to give an overall score representing the performance of the user.

CONTACTS AND LOCATIONS:
Overall Officials: Zahra Moussavi, Principal Investigator — University of Manitoba
Locations (1):
- Riverview Health Center, Winnipeg, Manitoba, Canada